CLINICAL TRIAL: NCT02035215
Title: Efficacy and Safety of Co-administration of Omacor Plus Atorvastatin Compared With Atorvastatin Monotherapy in Patients With Type Ⅱb Dyslipidemia: a Multicenter, Double-blind, Randomized, Active-controlled, Parallel, Phase Ⅲ Study
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Omega-3-acids Ethylesters 90 in Type Ⅱb Hyperlipidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-OM-8302
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Hyperlipidemia, Familial Combined
Keywords: Hyperlipidemia, Familial Combined; Omega 3 acids ethylesters 90; Atorvastatin
MeSH Terms: conditions — Hyperlipidemia, Familial Combined | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 20mg, Omega-3-acids ethylesters 90 4g (Experimental): Atorvastatin calcium 20mg, Omega-3-acids ethylesters 90 4g: po, q.d
  Interventions: Drug: Atorvastatin 20mg; Drug: Omega-3-acids ethylesters 90 4g
- Atorvastatin 20mg, Placebo (Placebo Comparator): Atorvastatin calcium 20mg, Placebo for Omega-3-acids ethylesters 90 4g: po, q.d
  Interventions: Drug: Atorvastatin 20mg; Other: Placebo(Omega-3-acids ethylesters 90)

INTERVENTIONS:
Drug: Atorvastatin 20mg
  Other Names: Lipitor 20mg
Drug: Omega-3-acids ethylesters 90 4g
  Other Names: Omacor Soft Capsule 4g
  Arms: Atorvastatin 20mg, Omega-3-acids ethylesters 90 4g
Other: Placebo(Omega-3-acids ethylesters 90)
  Arms: Atorvastatin 20mg, Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combination therapy of omega-3-acids ethylesters 90/Atorvastatin calcium in type Ⅱb hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* LDL≥160mg/dl, 200mg/dl≤TG<500mg/dl
* In the case of smokers, he agrees should be smoke-free
* In the case of women of childbearing age, urine pregnancy test must be negative

Exclusion Criteria:

* Patients with acute artery disease within 3 months
* History of revascularization procedure or aneurism operation within 6months
* Patients with myopathy, rhabdomyolysis
* Patients with pancreatitis
* Patients with HIV positive
* History of malignant tumor within 2 years
* Patients must be treated with medications prohibited for concomitant use during study period
* Patients with uncontrolled hypertension(SBP>180mmHg or DBP>110mmHg)
* Serum Creatinine>1.2mg/dl(female), >1.4mg/dl(male)
* AST or ALT > 2X ULN
* CPK > 2X ULN
* Patients with galactose intolerance or Lapp lactase deficiency, glucose-galactose malabsorption
* Allergy or Hypersensitive to investigational drug
* History of drug or alcohol abuse within 2 years
* In the case of smokers, who do not intend to non smoking
* Women with pregnant, breast-feeding
* Patients treated with any investigational drugs within 1 month at the time consents are obtained
* Not eligible to participate for the study at the discretion of investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The mean percent change of Triglyceride(TG) | from baseline at week 8

SECONDARY OUTCOMES:
The mean percent change of Triglyceride(TG) | from baseline at week 4
The mean percent change of Total Cholesterol(TC), LDL-C, HDL-C | from baseline at week 4,8

CONTACTS AND LOCATIONS:
Overall Officials: Hong Seog Seo, Ph.D., Principal Investigator — Korea University Guro Hospital; Hee Kyoung Cheon, Ph.D., Principal Investigator — Uijongbu St. Mary's Hospital; Sang-Ho Jo, Ph.d., Principal Investigator — Hallym University Medical Center; Mi-Seung Shin, Ph.D, Principal Investigator — Gachon University Gil Medical Center
Locations (4):
- South Korea (4):
  - Hallym University Sacred Heart Hospital, Anyang, Gyeonggi
  - Gachon University Gil Hospital, Incheon
  - Korea University Guro Hospital, Seoul
  - Uijongbu St. Mary's Hospital, Uijongbu, Gyeonggi